CLINICAL TRIAL: NCT06010199
Title: Risk Stratification Value of Biomarkers in Patients With Myocarditis (FORWARD): a National, Multicenter, Retrospective-prospective, Cohort Study
Brief Title: Risk Stratification Value of Biomarkers in Patients With Myocarditis
Acronym: FORWARD
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-169
Record Dates: First submitted 2023-07-06; First posted 2023-08-24 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-03

CONDITIONS: Myocarditis
Keywords: Myocarditis; Biomarker; Risk stratification
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood, urine, feces.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myocarditis group: All enrolled patients are administered antiviral drugs, glucocorticoids, immunoglobulins, and other standard treatments. Additionally, the decision to provide ECMO support therapy is based on the severity of the patient's condition.

SUMMARY:
The aim of this study is to collect clinical data and biological specimens from patients with myocarditis and construct a predictive model for the prognosis of myocarditis.

DETAILED DESCRIPTION:
The aim of this study is to retrospectively and prospectively collect clinical data and biological specimens from patients with myocarditis who meet the inclusion and exclusion criteria. General molecular biology analysis, genome sequencing, transcriptome sequencing, methylation sequencing, metabolomics analysis, proteomics analysis, genome-wide chromosome conformation capture and other techniques are used to construct a prognosis prediction model for myocarditis.

ELIGIBILITY:
Inclusion Criteria:

* All patients should meet the diagnostic criteria for myocarditis
* Patients who are regularly followed up at the corresponding cardiovascular center

Exclusion Criteria:

* Age <3 years or >80 years
* Pregnant or lactating women
* The patient refused to sign the informed consent and refused to participate in the study
* None of the above is consistent, but the patient cannot sign the informed consent temporarily due to coma and other reasons, and there is no legal representative to sign it instead. Depending on the condition, the patient may not wake up to sign the informed consent

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All hospitalized patients who meet the diagnostic criteria for myocarditis and undergo regular follow-up at the corresponding cardiovascular center are included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in the incidence of MACCE | 1, 3, 6 months after enrollment; and 1, 2, 3, 4, 5 years after enrollment.
  MACE (major adverse cardiovascular events) including all-cause death, myocardial infarction, stroke and coronary revascularization surgery. The MACCE will be assessed from the medical records.

SECONDARY OUTCOMES:
Change in the incidence of all-cause death | 1, 3, 6 months after enrollment; and 1, 2, 3, 4, 5 years after enrollment.
  All-cause death diagnosed by clinical doctors will be assessed from the medical records
Change in the incidence of myocardial infarction | 1, 3, 6 months after enrollment; and 1, 2, 3, 4, 5 years after enrollment.
  Myocardial infarction diagnosed by clinical doctors will be assessed from the medical records
Change in the incidence of stroke | 1, 3, 6 months after enrollment; and 1, 2, 3, 4, 5 years after enrollment.
  Stroke diagnosed by clinical doctors will be assessed from the medical records
Change in the incidence of coronary revascularization surgery | 1, 3, 6 months after enrollment; and 1, 2, 3, 4, 5 years after enrollment.
  Coronary revascularization surgery completed by clinical doctors will be assessed from the medical records

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yan, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; Guoliang Li, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China